CLINICAL TRIAL: NCT07258329
Title: Screening Della Compromissione Fetale Intrapartum Mediante Utilizzo Dei Marcatori Placentari
Brief Title: Screening for Intrapartum Fetal Compromise Using Placental Biomarkers
Status: Recruiting | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: PLGF_IFC
Record Dates: First submitted 2025-11-19; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Pregnant Women

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the association between placental markers (sFlt-1, PlGF, and the sFlt-1/PlGF ratio) and intrapartum fetal compromise, assessed on the basis of the cardiotocographic tracing.

DETAILED DESCRIPTION:
The development of placentation during pregnancy involves two simultaneous processes: the invasion of maternal spiral arteries by cytotrophoblasts and the branching of the fetal vascular tree. These mechanisms, regulated by factors such as VEGF, PlGF, sFlt-1, and PAPP-A, ensure an adequate supply of oxygen and nutrients to the fetus. When these processes are impaired, placental dysfunction develops, characterized by high vascular resistance, hypoperfusion, and oxidative stress, which can predispose to complications such as preeclampsia, fetal growth restriction, gestational diabetes, placental abruption, and preterm birth.

During labor, uterine contractions can reduce uteroplacental perfusion by up to 60%. A healthy fetus with a normally functioning placenta can tolerate these transient reductions through compensatory mechanisms, whereas a fetus with abnormal placentation may exhibit signs of compromise, such as abnormal heart rate patterns or the presence of meconium, and, in cases of severe hypoxia, may face more serious risks.

The clinical challenge is to identify, before labor, fetuses that, despite appropriate growth, have a placenta unable to withstand the stress of delivery. Some studies have investigated Doppler velocimetry, particularly the Cerebro-Placental Ratio, but its predictive ability at term is modest. The role of placental markers (PlGF, sFlt-1, sFlt-1/PlGF) in predicting intrapartum fetal compromise also remains uncertain, with conflicting results reported in the literature. Since these markers are altered in pregnancies with placental dysfunction, their combination with antenatal risk factors may allow better identification of fetuses at risk, guiding clinicians in labor management and the choice of delivery mode.

This study will enroll participants using a retrospective and prospective approach. The primary aim is to evaluate the association between placental markers and intrapartum fetal compromise based on cardiotocographic tracings. Secondary aims include assessing their relationship with fetal acidosis, low Apgar scores, and admission to the neonatal intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Gestational age ≥ 32 weeks
* Obtaining informed consent for participation in the study and for the processing of personal data
* Pregnant patients with an indication to perform placental marker testing as part of routine clinical practice
* Patients who will deliver at the Obstetrics Units of the participating centers

Exclusion Criteria:

- Absolute contraindications to vaginal delivery (placenta previa, vasa previa, placenta accreta, previous myomectomy)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: The study will enroll pregnant patients who present to the Obstetrics Units of the participating centers
Sampling Method: Non-Probability Sample
Enrollment: 428 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Diagnosed with Intrapartum Fetal Compromise Based on Cardiotocographic Tracing | At the time of delivery
  Association between placental markers and intrapartum fetal compromise

SECONDARY OUTCOMES:
Number of Participants With Fetal Acidosis (pH ≤ 7.0 or Base Excess ≥ -12) | At the time of delivery
  Association between placental markers and fetal acidosis
Number of Participants With 5-Minute Apgar Score < 7 | At the time of delivery
  Association between placental markers and low birth Apgar score
Number of Newborns Transferred to Neonatal Intensive Care Unit (NICU) for Birth-Related Hypoxia | At the time of delivery
  Association between placental markers and admission to the neonatal intensive care unit

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna
  - IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Milano